CLINICAL TRIAL: NCT01769183
Title: Topical Squalamine in the Treatment of Retinal Neovascularization From Proliferative Diabetic Retinopathy
Brief Title: Squalamine for the Treatment in Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elman Retina Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ohr-003
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Retinal Neovascularization
Keywords: Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Retinal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Squalamine (Experimental): Study eyes will be assigned to receive Squalamine. The dose will be one drop twice daily. If neovascularization fails to regress at week one or if neovascularization returns within the study, the dose will be increased to four times daily. In that case, a one day and one week visit will be added after increasing the dose. Patients will continue administering study drug until week 20.
  Interventions: Drug: Squalamine Lactate ophthalmic solution 0.2%

INTERVENTIONS:
Drug: Squalamine Lactate ophthalmic solution 0.2% — Patients will start with Squalamine one drop twice daily to the affected eye. If at one week the neovascularization shows no sign of regression, then the dose will be doubled to four times daily with a follow up at one day and one week following the increased dose frequency, then resuming the schedule at four weeks. If neovascularization returns within the study, the dose will be doubled to four times daily. In that case, a one day and one week visit will be added after increasing the dose. Squalamine treatment will discontinue after the week 20 visit.

SUMMARY:
The purpose of this study is to determine the efficacy in the use of topical Squalamine Lactate Ophthalmic Solution, 0.2% in the treatment of retinal neovascularization resulting from proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Individuals <18 years old are not being included because PDR is so rare in this age group that the diagnosis of PDR may be questionable.
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Any one of the following will be considered to be sufficient evidence that diabetes is present:
* Current regular use of insulin for the treatment of diabetes
* Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
* Documented diabetes by ADA and/or WHO criteria (see Procedures Manual for definitions)
* At least one eye meets the study eye criteria
* Able and willing provide informed consent

Exclusion Criteria:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Individuals in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.
* Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied.
* Note: study participants cannot receive another investigational drug while participating in the study.
* Known allergy to any component of the study drug.
* Blood pressure > 180/110 (systolic above 180 or diastolic above 110).
* If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
* Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization.
* These drugs should not be used during the study.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.
* Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
* Individual is expecting to move out of the area of the clinical center during the study.
* History of allergy to Squalamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Proportion with complete regression of neovascularization on fundus photography at one month | 1 Month

SECONDARY OUTCOMES:
Mean Change in Visual Acuity from Baseline to 5 Months | 5 months

OTHER OUTCOMES:
Proportion with partial regression of neovascularization on fundus photography | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Elman Retina Group, P.A., Baltimore, Maryland, United States